CLINICAL TRIAL: NCT07135076
Title: PARodontitis And Type 2 DIabetes in Elderly Subjects
Acronym: PARADIES
Status: Completed | Type: Observational
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Praxis am Posthof, Hameln, Germany (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director of Department of Clinical Nutrition, German Institute of Human Nutrition
Other Study IDs: PARADIES
Record Dates: First submitted 2020-07-21; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2020-07

CONDITIONS: Parodontitis; Type2 Diabetes
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- type 2 diabetes: patients are examined for symptoms (questionnaire) and clinical signs of parodontitis (PSI), data from the individual dentists are collected, too

SUMMARY:
PARADIES is a cross-sectional observational study on Parodontitis and Type-2-diabetes. Its purpose is to collect data on the prevalence of Parodontitis and Type-2-diabetes in a regular out-patient setting, to provide insight into predictive conditions (such as comorbidities, blood parameters, clinical symptoms etc.)

DETAILED DESCRIPTION:
PARADIES is a cross-sectional observational study on Parodontitis and Type-2-diabetes. Its purpose is to collect data on the prevalence of Parodontitis and Type-2-diabetes in a regular out-patient setting, to provide insight into predictive conditions (such as comorbidities, blood parameters, clinical symptoms etc.).

Data is collected once only, includes questionnaires on dental symptoms and dental condition, dental hygiene, general clinical anamnesis, recent state of routine blood parameters and medication.

ELIGIBILITY:
Inclusion Criteria:

* type-2-diabetes

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type-2-diabetes patients from an out-patient endocrinologist in Hameln, Germany
Sampling Method: Non-Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Survey on prevalence of confirmed and assumed parodontitis / parodontitis stages, stratified by type of diabetes and sex | baseline
  prevalence of confirmed and assumed parodontitis / parodontitis stages, stratified by type of diabetes and sex
Survey on co-prevalence of confirmed / assumed parodontitis / parodontitis stages with hypertension, depression and diabetic microvascular complications | baseline
  co-prevalence of confirmed / assumed parodontitis / parodontitis stages with hypertension, depression and diabetic microvascular complications
Questionnaire on prediction analysis on prevalence of confirmed and assumed parodontitis / parodontitis stages | baseline
  prediction analysis on prevalence of parodontitis / parodontitis stages based on type of diabetes, diabetes duration / diabetes onset, sex, co-morbidities, metabolic state (BMI, fasting glucose, HbA1c, diabetes medication), smoking, dental hygiene and compliance, quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg
  - DIfE (German Institute for Human Nutrition), Berlin

IPD SHARING:
Plan to Share IPD: No